CLINICAL TRIAL: NCT03835065
Title: Long Arm Vs Short Arm Fiberglass Cast for Treatment of Displaced Distal Radius Fractures: A Multi-Center Randomized Control Trial
Brief Title: Long Arm Vs Short Arm Fiberglass Cast for Treatment of Displaced Distal Radius Fractures
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study expired on 2/11/2025.
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-1930
Record Dates: First submitted 2018-11-14; First posted 2019-02-08 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2024-03

CONDITIONS: Distal Forearm Fractures
Keywords: Displaced distal third forearm; Pediatric Patients; Closed reduction; Cast; Patient centered outcome data; RCT
MeSH Terms: conditions — Wrist Fractures | interventions — Closed Fracture Reduction

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Long Arm Fiberglass Cast (Active Comparator): Conscious sedation will be provided to patient while the reduction is performed by a cast trained orthopedic resident using standard techniques under fluoroscopic guidance. The arm will be held by an assistant or finger traps in the absence thereof. The arm will not be suspended until after the manipulation is performed. A stockingette and webril will first be applied, after which the short arm fiberglass portion of the cast will be applied. After short arm casting has been appropriately placed, randomization group will be revealed. Casting will be extended to the shoulder joint if the patient is assigned to the long arm cast group. The mold will then be applied and cast construct will be bivalved and taped.
  Interventions: Procedure: Closed Reduction; Other: Long Arm Fiberglass Cast
- Short Arm Fiberglass Cast (Experimental): Conscious sedation will be provided to patient while the reduction is performed by a cast trained orthopedic resident using standard techniques under fluoroscopic guidance. The arm will be held by an assistant or finger traps in the absence thereof. The arm will not be suspended until after the manipulation is performed. A stockingette and webril will first be applied, after which the short arm fiberglass portion of the cast will be applied. After short arm casting has been appropriately placed, randomization group will be revealed. Casting will be complete at this point if the patient is assigned to the short arm cast group. The mold will then be applied and cast construct will be bivalved and taped.
  Interventions: Procedure: Closed Reduction; Other: Short Arm Fiberglass Cast

INTERVENTIONS:
Procedure: Closed Reduction — The primary goal of closed reduction is to maintain appropriate bony alignment and angulation to allow for appropriate healing.
Other: Long Arm Fiberglass Cast — A stockingette and webril will first be applied, after which the short arm fiberglass portion of the cast will be applied. After short arm casting has been appropriately placed, randomization group will be revealed. Casting will be extended to the shoulder joint if the patient is assigned to the long arm cast group. The mold will then be applied and cast construct will be bivalved and taped.
  Arms: Long Arm Fiberglass Cast
Other: Short Arm Fiberglass Cast — A stockingette and webril will first be applied, after which the short arm fiberglass portion of the cast will be applied. After short arm casting has been appropriately placed, randomization group will be revealed. Casting will be complete at this point if the patient is assigned to the short arm cast group. The mold will then be applied and cast construct will be bivalved and taped.
  Arms: Short Arm Fiberglass Cast

SUMMARY:
The aim of the study is to determine by multicenter randomized controlled trial whether short arm fiberglass casts are as effective as long arm casts for immobilizing displaced pediatric distal third forearm fractures that have undergone closed reduction.

The primary outcome is loss of reduction requiring cast wedging, recasting, repeat reduction, or surgical intervention.

Secondary outcomes will include Patient Reported Outcome Measures for physical function, such as Pedi-FABS, PROMIS (Patient Reported Outcomes Measurement Information System) Upper Extremities , and UCLA (University of California Los Angelos) Activity Scale, and pain/comfort levels,such as PROMIS Pediatric Pain Interference, PROMIS Pediatric Pain Intensity, and VAS ( Visual Analogue Scale) comfort in cast. In addition, secondary outcomes include complications (skin irritation, compartment syndrome, elbow stiffness, cast saw burns etc). The investigators will assess potential risk factors for loss of reduction including initial displacement, level of fracture (physeal, metaphyseal, meta-diaphyseal), initial translation, initial angulation, age, sex, cast index, padding index, adequacy of initial reduction, and provider level of training.

DETAILED DESCRIPTION:
The most common type of fracture in pediatric patients is the distal third forearm fracture, with over 600,000 cases in the in the United States each year. Traditionally long arm casts have been used for displaced distal forearm fractures, but it may be the case that short arm casts are sufficient. Three RCTs (Randomized Control Trials) have been performed comparing the efficacy of plaster short and long arm casts for displaced distal forearm fractures; these studies have shown no significant difference in angulation or displacement. If short and long arm casts offer comparable stability, the short arm version would likely be desirable as patient satisfaction and cost effectiveness are improved with short arm casts.

Despite the results of three well-executed RCTs, it is still common practice for long arm casts to be applied for distal forearm fractures. Many surgeons continue to recommend that their residents apply long arm casts for all displaced forearm fractures, including distal third fractures. At NYP (New York Presbyterian) Cornell and NYP Queens, residents routinely apply long arm casts for all forearm fractures.

Long arm casts are more likely to result in elbow stiffness, although this is often a temporary complication. Long arm casts also require more material and take longer to apply or remove, potentially leading to higher treatment costs. Additionally, when a longer cast is worn there is a larger distance where a cast burn could occur. Skin irritation, particularly at the cubital fossa, is likely more common with a long arm cast, and they are overall less comfortable, due to elbow restriction and a heavier weight.

Short arm casts that are well molded to the arm's contours have been shown to control forearm supination and pronation. A low cast index has been shown to significantly increase the rate of fracture redisplacement. The cast index determines the quality of cast molding, and is measured by dividing the sagittal width of the cast by the coronal width. Substantial changes in cast angulation have been attributed to poor cast-molding and a low cast index. The results suggested that short arm casts when appropriately molded can be effective in treating fractures of the distal third of the forearm.

If short arm casts are equivalent in providing stability for distal third forearm fractures, providers should be using them preferentially to avoid the potential complications of elbow stiffness, cast burn, skin irritation, and patient dissatisfaction. However, surgeons persist with using long arm casts. Rationale for the persistent use of long arm cast is believed to include anecdotal concerns of residents placing inadequate short arm casts, leading to an increased risk for translation or angulation requiring recasting.

Previous RCTs, however, do not provide clear recommendations, merely demonstrating that treatment using short and long arm casts lead to similar outcomes. Additionally, these past RCTs have limitations. Previous studies were conducted with plaster casts and could not extend their findings to other casting material. Valving techniques were also not noted in these studies; it is unclear whether or not casts were bivalved, which is currently the standard of care in the United States. These previous studies also randomized patients to short or long arm cast prior to cast application. As a result, it is possible that when long arm casts were applied the portion of cast overlying the fracture site was not molded as carefully as for short arm casts. Previous studies commented on cast index, but it was not clear whether residents were trained in ideal cast application and molding prior to study initiation. Finally, the outcome measures used in previous studies were an arbitrary loss in angulation or translation, instead of a focus on whether the fracture slipped sufficiently to change the treatment required (need for cast wedging, repeat reduction and casting, or surgical intervention).

The aim of the study is to determine by multicenter randomized controlled trial whether short arm fiberglass casts are as effective as long arm casts for immobilizing displaced pediatric distal third forearm fractures that have undergone closed reduction.

ELIGIBILITY:
Inclusion Criteria:

Patients 4-12 years of age

* Displaced distal third forearm fracture (physeal, metaphyseal, meta-diaphyseal) requiring closed reduction
* Displacement must be: For children 4-9: angulation >30 degrees and/or 100% translation on either AP (anteroposterior) or lateral view. For children 10-12: angulation > 15 degrees and/or >50% translation on either AP or lateral view

Exclusion Criteria:

* Patients undergoing additional orthopedic procedures at the time closed reduction of distal arm fracture
* Patient with a presenting open fracture
* A known pathologic fracture
* Patient with a refracture through pre-existing fracture lines
* Patients with compartment syndrome or neuropathy

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2019-02-12 (Actual); Primary Completion 2025-02-11 (Actual); Study Completion 2025-02-11 (Actual)

PRIMARY OUTCOMES:
Patients requiring repeat intervention due to loss of alignment | Up to 7 months
  Proportion of patients requiring repeat intervention (cast wedging, recasting, or surgical intervention) following short arm vs long arm cast application.

SECONDARY OUTCOMES:
Pain assessed by patient reported outcomes - Surveys | 1 week +/- 5 days visit, 3 weeks +/- 1 week, 6 weeks +/- 1 week, 3 months +/- 2 weeks , 6 months +/- 4 weeks
  Patient Reported Outcome Measures for pain as assessed by PROMIS(Patient-Reported Outcomes Measurement Information System) Pediatric Pain Interference. Highest raw score is 32, lowest raw score is 0, it is interpreted by t-score.
Pain assessed by patient reported outcomes - Surveys | 1 week +/- 5 days visit, 3 weeks +/- 1 week, 6 weeks +/- 1 week, 3 months +/- 2 weeks , 6 months +/- 4 weeks
  Patient Reported Outcome Measures for pain as assessed by PROMIS (Patient-Reported Outcomes Measurement Information System) Pediatric Pain Intensity. Highest raw score is 32, lowest raw score is 0, it is interpreted by t-score.
Comfort assessed by patient reported outcomes - Scale | 1 week +/- 5 days visit, 3 weeks +/- 1 week, 6 weeks +/- 1 week, 3 months +/- 2 weeks , 6 months +/- 4 weeks
  Patient Reported Outcome Measures for pain as assessed by Visual Analog Scale (VAS) comfort in cast. VAS measures the amount of pain that a patient feels currently and ranges across a continuum from none to an extreme amount of pain. Higher values represent more pain/ worse outcome.
Physical function assessed by patient reported outcomes - Surveys | 1 week +/- 5 days visit, 3 weeks +/- 1 week, 6 weeks +/- 1 week, 3 months +/- 2 weeks , 6 months +/- 4 weeks
  Patient Reported Outcome Measures for pain as assessed by Pedi-FABS ( Pediatric Functional Activity Brief Scale). Scoring of the Hospital for Special Surgery PediatricFunctional Activity Brief Scale is performed by addingpoints from each question for total possible score range from1 to 30 points. For ''Running'', ''Cutting'', ''Decelerating'',''Pivoting'', ''Duration'', and ''Endurance'', each question is worth 0, 1, 2, 3, or 4 points. Higher values mean that the child is more active.
Physical function assessed by patient reported outcomes - Surveys | 1 week +/- 5 days visit, 3 weeks +/- 1 week, 6 weeks +/- 1 week, 3 months +/- 2 weeks , 6 months +/- 4 weeks
  Patient Reported Outcome Measures for pain as assessed by PROMIS ( Patient-Reported Outcomes Measurement Information System) Upper Extremity. Within the Pediatric Upper Extremity short form, there are two items (3880R2 and 3881R1) with collapsed response categories. These items have response options scored as 3=With no trouble, 2=With a little trouble, 1=With some trouble, 0=With a lot of trouble, 0=Not able to do.
Physical function assessed by patient reported outcomes - Surveys | 1 week +/- 5 days visit, 3 weeks +/- 1 week, 6 weeks +/- 1 week, 3 months +/- 2 weeks , 6 months +/- 4 weeks
  Patient Reported Outcome Measures for pain as assessed by UCLA Activity Scale (University of California, Los Angeles Activity Scale). 1 is the lowest raw score, and 10 is the highest raw score. 1= 1: Wholly Inactive, dependent on others, and can not leave residence and 10= 10: Regularly participates in impact sports.
Number of Participants with complications | 1 week +/- 5 days visit, 3 weeks +/- 1 week, 6 weeks +/- 1 week, 3 months +/- 2 weeks , 6 months +/- 4 weeks
  irritation, compartment syndrome, elbow stiffness, cast saw burns etc

CONTACTS AND LOCATIONS:
Overall Officials: Emiyl R Dodwell, MD MPH FRCSC, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nellans KW, Kowalski E, Chung KC. The epidemiology of distal radius fractures. Hand Clin. 2012 May;28(2):113-25. doi: 10.1016/j.hcl.2012.02.001. Epub 2012 Apr 14. PMID 22554654
- [Background] Bohm ER, Bubbar V, Yong Hing K, Dzus A. Above and below-the-elbow plaster casts for distal forearm fractures in children. A randomized controlled trial. J Bone Joint Surg Am. 2006 Jan;88(1):1-8. doi: 10.2106/JBJS.E.00320. PMID 16391243
- [Background] Webb GR, Galpin RD, Armstrong DG. Comparison of short and long arm plaster casts for displaced fractures in the distal third of the forearm in children. J Bone Joint Surg Am. 2006 Jan;88(1):9-17. doi: 10.2106/JBJS.E.00131. PMID 16391244
- [Background] Paneru SR, Rijal R, Shrestha BP, Nepal P, Khanal GP, Karn NK, Singh MP, Rai P. Randomized controlled trial comparing above- and below-elbow plaster casts for distal forearm fractures in children. J Child Orthop. 2010 Jun;4(3):233-7. doi: 10.1007/s11832-010-0250-1. Epub 2010 Mar 17. PMID 21629372
- [Background] Colaris JW, Allema JH, Biter LU, Reijman M, van de Ven CP, de Vries MR, Bloem RM, Kerver AJ, Verhaar JA. Conversion to below-elbow cast after 3 weeks is safe for diaphyseal both-bone forearm fractures in children. Acta Orthop. 2013 Oct;84(5):489-94. doi: 10.3109/17453674.2013.850010. Epub 2013 Oct 31. PMID 24171685
- [Background] Worlock P, Stower M. Fracture patterns in Nottingham children. J Pediatr Orthop. 1986 Nov-Dec;6(6):656-60. doi: 10.1097/01241398-198611000-00003. PMID 3793885
- [Background] Webb JE, Lewallen LW, Christophersen C, Krych AJ, McIntosh AL. Clinical outcome of internal fixation of unstable juvenile osteochondritis dissecans lesions of the knee. Orthopedics. 2013 Nov;36(11):e1444-9. doi: 10.3928/01477447-20131021-30. PMID 24200451
- [Background] Kamat AS, Pierse N, Devane P, Mutimer J, Horne G. Redefining the cast index: the optimum technique to reduce redisplacement in pediatric distal forearm fractures. J Pediatr Orthop. 2012 Dec;32(8):787-91. doi: 10.1097/BPO.0b013e318272474d. PMID 23147621
- [Background] Chess DG, Hyndman JC, Leahey JL, Brown DC, Sinclair AM. Short arm plaster cast for distal pediatric forearm fractures. J Pediatr Orthop. 1994 Mar-Apr;14(2):211-3. doi: 10.1097/01241398-199403000-00015. PMID 8188836